CLINICAL TRIAL: NCT01069874
Title: Cluster-randomised, Double-Blind, Placebo-Controlled Trial of Vitamin D Supplementation for the Prevention of Influenza and Other Respiratory Infections in Sheltered Accommodation (ViDiFlu)
Brief Title: Trial of Vitamin D Supplementation for the Prevention of Influenza and Other Respiratory Infections (ViDiFlu)
Acronym: ViDiFlu
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: National Health Service, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2009-010085-35
Record Dates: First submitted 2010-02-16; First posted 2010-02-17 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-02

CONDITIONS: Respiratory Tract Infections; Influenza
Keywords: Bone Density Conservation Agents; Cholecalciferol; Communicable Diseases; Growth Substances; Housing for the Elderly; Infection; Micronutrients; Pharmacologic Actions; Physiological Effects of Drugs; Respiratory Tract Diseases; Vitamins; Respiratory Tract Infections/prevention & control*; Vitamin D
MeSH Terms: conditions — Respiratory Tract Infections; Influenza, Human; Communicable Diseases; Infections; Respiratory Tract Diseases | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Miglyol oil (Placebo Comparator): Miglyol oil will be administered in 2-monthly oral bolus doses over a period of one year
  Interventions: Dietary Supplement: Miglyol oil
- Vigantol oil (Active Comparator): Vigantol oil will be administered in 2-monthly oral bolus doses over a period of one year
  Interventions: Dietary Supplement: Cholecalciferol (Vitamin D/Vigantol oil)

INTERVENTIONS:
Dietary Supplement: Cholecalciferol (Vitamin D/Vigantol oil) — Cholecalciferol will be administered as 2-monthly oral bolus doses of Vigantol oil over a period of one year
  Other Names: Vigantol oil
  Arms: Vigantol oil
Dietary Supplement: Miglyol oil — Miglyol oil will be administered as 2-monthly oral bolus doses of Miglyol oil over a period of one year
  Arms: Miglyol oil

SUMMARY:
Purpose: The study null hypothesis is that vitamin D supplementation will not influence time to acute respiratory tract infection in sheltered accommodation residents.

DETAILED DESCRIPTION:
The study population will comprise sheltered accommodation residents and staff fulfilling eligibility criteria. Half of the sheltered accommodation schemes will be randomly allocated to 2-monthly oral bolus vitamin D supplementation (Vigantol oil) over a period of one year, and half to placebo.

Participants will be followed for one year.

ELIGIBILITY:
Inclusion Criteria:

* Permanent resident or member of staff at sheltered accommodation unit
* If a woman of child-bearing potential, is sexually abstinent or has negative pregnancy test within 7 days of recruitment and agrees to use reliable form of contraception until she has completed the study
* Able to give written informed consent to participate
* Age ≥ 16 years on day of first dose of IMP

Exclusion Criteria:

* Current diagnosis of asthma or chronic obstructive pulmonary disease
* Chronic upper or lower respiratory infection or other condition causing chronic cough
* Condition requiring treatment with vitamin D at a dose of > 10 micrograms vitamin D/day
* Episode of upper or lower respiratory tract infection up to 28 days before first dose of IMP
* Known sarcoidosis, hyperparathyroidism, nephrolithiasis, active tuberculosis, vitamin D intolerance, liver failure, renal failure, terminal illness, lymphoma or other malignancy not in remission at time of recruitment
* Taking benzothiadiazine derivative, cardiac glycoside, carbamazepine, phenobarbital, phenytoin, primidone or long-term immunosuppressant therapy
* Taking oral preparation containing > 10 micrograms vitamin D/day up to 2 months before first dose of IMP
* Using topical vitamin D analogue
* Treatment with any investigational medical product or device up to 4 months before first dose of IMP
* Breastfeeding, pregnant or planning a pregnancy
* Baseline corrected serum calcium > 2.65 mmol/L
* Baseline serum creatinine > 125 micromol/L
* Inability to complete symptom diary with / without assistance
* Cognitive impairment or communication problem precluding informed consent or successful completion of study evaluations

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2010-03; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Time to first respiratory tract infection (upper or lower) in sheltered accommodation residents | One year

SECONDARY OUTCOMES:
Time to first respiratory tract infection (upper or lower) in sheltered accommodation staff | One year
Annual rate of episodes of upper / lower respiratory infection in sheltered accommodation residents / staff | One year
Time to unscheduled health service use for respiratory tract infection in sheltered accommodation residents / staff | One year
Proportion of participants experiencing hypercalcaemia | One year

CONTACTS AND LOCATIONS:
Overall Officials: Adrian R Martineau, MRCP, Study Director — Queen Mary University of London
Locations (2):
- United Kingdom (2):
  - Hanover in Hackney Housing Association, London
  - Sanctuary Group Housing Association, London

REFERENCES:
- [Derived] Martineau AR, Hanifa Y, Witt KD, Barnes NC, Hooper RL, Patel M, Stevens N, Enayat Z, Balayah Z, Syed A, Knight A, Jolliffe DA, Greiller CL, McLaughlin D, Venton TR, Rowe M, Timms PM, Clark D, Sadique Z, Eldridge SM, Griffiths CJ. Double-blind randomised controlled trial of vitamin D3 supplementation for the prevention of acute respiratory infection in older adults and their carers (ViDiFlu). Thorax. 2015 Oct;70(10):953-60. doi: 10.1136/thoraxjnl-2015-206996. Epub 2015 Jun 10. PMID 26063508